CLINICAL TRIAL: NCT06441474
Title: Understanding and Addressing Rejection of Personalized Cancer Risk Information
Brief Title: Understanding and Addressing Rejection of Personalized Breast Cancer Risk Information in Women
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Cancer Institute (NCI) (NIH); National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 23-0345.cc; 1R01CA279953-01 (NIH)
Record Dates: First submitted 2024-05-22; First posted 2024-06-04 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Breast Cancer Female
Keywords: Risk rejection; Screening behaviour

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Breast cancer risk (Other): All participants receive a personal breast cancer risk estimate using the Gail Model
  Interventions: Behavioral: Presentation of personal breast cancer risk estimate

INTERVENTIONS:
Behavioral: Presentation of personal breast cancer risk estimate — All participants will be presented with their personal breast cancer risk estimate, calculated using the Gail Model

SUMMARY:
The Understanding and Addressing Rejection of Personalized Cancer Risk Information study is a longitudinal study conducted to understand the nature of phenomenon of personalized cancer risk rejection in the context of mammography screening.

DETAILED DESCRIPTION:
The Understanding and Addressing Rejection of Personalized Cancer Risk Information study seeks to understand the nature of the phenomenon of personalized cancer risk rejection in the context of mammography screening by 1) identifying demographic and psychological factors associated with risk rejection and 2) identify how risk rejection influences risk-concordant mammography screening behavior. The study will test a priori theory-derived hypotheses about the precursors of risk rejection and the influence of rejection on real-life screening decision making.

The Breast Cancer Risk Assessment Tool (BCRAT) will be used to asses participant's breast cancer risk. This model is designed to estimate breast cancer risk in women 35-84, and uses the following predictors: 1) age, 2) age at first menstrual period, 3) age at first live birth, 4) first-degree relatives with breast cancer, 5) previous breast biopsy with atypical hyperplasia, and 6) race/ethnicity. Participants will be required to complete the baseline survey in which they receive their BCRAT model risk estimate and respond to that risk estimate. They will then complete a 12-month follow-up survey.

ELIGIBILITY:
Inclusion Criteria:

1. Female sex
2. Age 39-74 (i.e., people who are eligible for routine breast cancer screening and for whom guidelines recommend an informed, risk-based decision)
3. English literacy

Exclusion Criteria:

1. Prior diagnosis of

1. breast cancer
2. Ductal carcinoma in situ (DCIS)
3. Lobular carcinoma in situ (LCIS)
4. Known BRCA1/2 gene mutation
5. Cowan syndrome
6. Li-Fraumeni syndrome
7. Having received previous chest radiation for treatment of Hodgkin's lymphoma.

Ages: 39 Years to 74 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 750 (Estimated)
Dates: Start 2025-04-02 (Actual); Primary Completion 2027-04-02 (Estimated); Study Completion 2028-04-02 (Estimated)

PRIMARY OUTCOMES:
Risk rejection as measured by a numeric estimate. | At baseline survey
  Participants are asked whether they agree or disagree with their Gail Model risk estimate. An open text box allows them to write the risk number that they believe is accurate for them.
Risk-concordant information seeking | At baseline survey
  Participants will be given the opportunity to get more information about breast cancer screening, and will be given response options to receive information for women at lower than average risk, higher than average risk, or women with risk that is "about the same as a typical woman". Concordance is measured by agreement between the participants' actual risk estimate and the option that they choose.
Screening intentions | At baseline survey
  Participants are asked their plans to get a mammogram in the next 12 months. The question is answered on a 5-point will-will not Likert scale.

SECONDARY OUTCOMES:
Goldilocks Risk Skepticism | At baseline survey
  Participants are asked whether they think their personal breast cancer risk estimate provided by the Risk Calculator is: '1=Much too low', '2=A little too low', '3=Just right', '4=A little too high', '5=Much too high.' This variable will be treated as continuous in analysis, with values on either end of the range (i.e., closer to 1 or closer to 5) indicating higher risk skepticism.
Risk rejection as measured by a validated believability scale | At baseline survey
  4 questions will be asked to assess whether participants find their risk estimate to be believable. Those questions will be averaged to create a summary score. The questions are:
  1. Overall, how much do you agree or disagree with your personal breast cancer risk estimate?
  2. In my opinion, my personal breast cancer risk estimate was believable.
  3. In my opinion, my personal breast cancer risk estimate was convincing.
  4. In my opinion, my personal breast cancer risk estimate was accurate.
  Each question is answered on a 5-point agree-disagree Likert scale.
Risk rejection as measured by risk relative to a typical woman their age. | At baseline survey
  Participants are told their breast cancer risk compared to a typical woman their age. They are asked whether they agree or disagree with this information, and are given the following response options:
  1. I think my risk is higher than a typical woman my age.
  2. I think my risk is about the same as a typical woman my age.
  3. I think my risk is lower than a typical woman my age.
Participant score on Subjective numeracy | At baseline survey
  Based on the McNaughton et al. MDM 2015 study, participants are asked questions to assess how they think about numbers and how this may affect their opinions about their breast cancer risk estimate. These questions are:
  1. How good are you at working with fractions?
  2. How good are you at figuring out how much a shirt will cost if it is 25% off?
  3. How often do you find numerical information to be useful?
Participant score on Risk Comprehension | At baseline survey
  We will be measuring participants' judgement of risk comparisons by asking two questions on 'Which amount is bigger?'
  Response options for question 1 are:
  1. The participant's breast cancer risk out of 1,000 people
  2. 15 out of 1,000 people
  3. They are the same Response options for question 2 are
  1- The participant's cancer risk out of 1,000 2- 6 out of 100 3- They are the same
  Each item will be scored (binary) for correctness.

OTHER OUTCOMES:
Number of Participants who engage in additional breast cancer seeking behavior | At 12 month follow-up
  Participants are asked if they talked to a health provider about their breast cancer risk and/or received additional breast health services.
Participant score on Health literacy | At baseline survey
  Adapted from HINTS 4 Cycle 2, participants are asked questions on their perceived confidence in understanding and using health information. These questions are:
  1. How confident are you that you could find advice or information about your health if you needed it?
  2. How confident are you about your ability to take good care of your health?
  3. How confident are you about your ability to understand information about your health? Each questions is measured on a 5-point not all confident-completely confident Likert scale.
Receipt of screening | At 12 month follow-up survey
  Participants are asked if they received a mammogram in the past 12 months following the baseline survey.
Racial demographic of participants | At baseline survey
  Participants are asked about their race and whether or not they are of Hispanic or Latino origin.

CONTACTS AND LOCATIONS:
Overall Officials: Laura Scherer, PhD, Principal Investigator — University of Colorado, Denver; Erika Waters, PhD, Principal Investigator — Washington University at St. Louis
Locations (2):
- United States (2):
  - University of Colorado Denver, Aurora, Colorado
  - Washington University in St. Louis, St Louis, Missouri

IPD SHARING:
Plan to Share IPD: Yes
We will share di-identified data
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: We will share data and supporting information when we submit the first manuscript for publication.
Access Criteria: Anyone can access on the Open Science Framework
URL: https://osf.io